CLINICAL TRIAL: NCT04624971
Title: A Novel Prognostic Model of NPI for Risk-Predicting and Clinical Decision-making in Diffuse Large B-Cell Lymphoma in the Rituximab Era
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Other Study IDs: B2020-235-01
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the predictive value of a model of Nomogram Prognostic Index (NPI) in patients with Diffuse Large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of CD20+ DLBCL

Exclusion Criteria:

* primary central nervous system lymphoma
* "double-hit" lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with clinical information available
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5-year

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University,, Guangzhou
  - Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University,, Guangzhou